CLINICAL TRIAL: NCT00979836
Title: Randomized, Double-blind Multicenter Clinical Trial Comparing the Efficacy of Calcium Dobesilate With Placebo in the Treatment of Ulcer Secondaries to Chronic Venous Disease
Brief Title: Calcium Dobesilate for Chronic Venous Wounds
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The financial support was withdrawn.
Sponsor: Fundacion Iberoamericana Itaca (Other)
Collaborators: Esteve Pharmaceuticals, S.A. (Industry)
Responsible Party: Mª JOSÉ MARTINEZ ZAPATA, Centro Cochrane Iberoamericano
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-002858-37
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Ulcer
Keywords: venous; ulcer; phlebotonic; calcium dobesilate; clinical trial
MeSH Terms: conditions — Ulcer | interventions — Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium Dobesilate (Experimental)
  Interventions: Drug: Calcium Dobesilate
- Placebo (Placebo Comparator): The placebo is a capsule with the same presence of experimental drug.
  Interventions: Drug: Calcium Dobesilate

INTERVENTIONS:
Drug: Calcium Dobesilate — 500 mg/ three times/day for 6 months (capsules)
  Other Names: Doxium

SUMMARY:
The objective of the study is to assess the efficacy of calcium dobesilate for treating chronic venous wounds.

The hypothesis is that venous ulcers treated with standards measures (compressive measures) and calcium dobesilate will heal-up better than venous ulcers treated with standards measures (compressive measures) and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with venous ulcer (CEAP 6) that affect epidermis, dermis and/or subcutaneous tissue, with and area superior to 3 cm2
* Ankle-arm index 0.9 or superior
* Written informed consent of the patients

Exclusion Criteria:

* Patients with venous ulcer (CEAP 6) that affect bone or with and area inferior to 3 cm2
* Ankle-arm index inferior to 0.9
* No written informed consent of the patients
* Diabetes mellitus I y II
* Patients with renal failure and dialysis
* Vascular surgery needed
* Impossibility to use compressive measures on the leg
* Use of topic antibiotics, silver dressing, growth factors, plasma-rich in platelets, skin graft, pentoxifylline, ultrasounds, laser, hyperbaric oxygen, electric stimulation o vacuum.
* Pregnancy
* Breast feeding
* No anticonceptives measures
* Allergy or intolerance to phebotonics
* Background of neutropenia or leucopenia
* Basal leucocytes < 3.500/ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Healed venous ulcers | at 6 months of treatment

SECONDARY OUTCOMES:
Percentage of re-epithelization area (cm2) | at 6 month of treatment
Length of time to heal ulcers | during all the period of the study (12 months)
Ulcer recurrence | at 12 month
Ulcer pain | at 6 and 12 months
Safety | during the study (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Moreno Carriles, Rosa Mª, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (42):
- Spain (42):
  - Hospital General de Albacete, Albacete, Albacete
  - Hospital Germans Tries i Pujol, Badalona, Barcelona
  - CAP Joanic, Barcelona, Barcelona
  - Hospital Sant Jaume de Calella, Calella, Barcelona
  - CAP El Castell, Castelldefels, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Consorci Hospitalari de Mataró, Mataró, Barcelona
  - CAP Pineda de Mar, Pineda de Mar, Barcelona
  - Corpotació Sanitària Parc Taulí, Sabadell, Barcelona
  - CAP Sitges, Sitges, Barcelona
  - CAP El Remei, Vic, Barcelona
  - Hospital de Vic, Vic, Barcelona
  - CAP Doctor Guillermo Masriera i Guardiola, Vilassar de Mar, Barcelona
  - CAP Les Corts, Barcelona, Catalonia
  - CAP Gaudí, Barcelona, Catalonia
  - CAP Sagrada Familia, Barcelona, Catalonia
  - CAP Vila de Gràcia, Barcelona, Catalonia
  - EAP Sardenya, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Dos de Maig, Barcelona, Catalonia
  - CAP la Sagrera, Barcelona, Catalonia
  - CAPSE, Barcelona, Catalonia
  - ABS Encants, Barcelona, Catalonia
  - ABS Lesseps, Barcelona, Catalonia
  - CAP la Salut, Barcelona, Catalonia
  - CAP Barceloneta, Barcelona, Catalonia
  - CAP Vila Olímpica, Barcelona, Catalonia
  - CAP Albera Salut, Peralada, Girona
  - Hospital de Leon, León, Leon
  - Fundación Hospital de Alcorcón, Alcorcón, Madrid
  - Hospital de Getafe, Getafe, Madrid
  - Complejo Hospitalario de Son Dureta, Mallorca, Mallorca
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - CAP Vila-Rodona, Vilarrodona, Tarragona
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital Platon, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital San Pedro de Logroño, Logroño
  - Hospital la Princesa, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid

REFERENCES:
- [Derived] Martinez-Zapata MJ, Vernooij RW, Simancas-Racines D, Uriona Tuma SM, Stein AT, Moreno Carriles RMM, Vargas E, Bonfill Cosp X. Phlebotonics for venous insufficiency. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD003229. doi: 10.1002/14651858.CD003229.pub4. PMID 33141449